CLINICAL TRIAL: NCT07269600
Title: The Effects of Sarcopenia on Cervical Proprioception, Kinesiophobia and Pressure Pain Threshold in Geriatric Nursing Home Residents
Brief Title: Effects of Sarcopenia on Proprioception, Kinesiophobia, and Pressure Pain Threshold
Status: Active, not recruiting | Type: Observational
Sponsor: Atılım University (Other)
Responsible Party: Principal Investigator, Beyza Doğanbaz, pyhsiotherapist, Atılım University
Other Study IDs: Beyza-ftr-01
Record Dates: First submitted 2024-11-14; First posted 2025-12-08 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-03

CONDITIONS: Sarcopenia in Elderly
Keywords: Pressure pain threshold; sarcopenia; crevical proprioception; kinesiophobia
MeSH Terms: conditions — Sarcopenia; Kinesiophobia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 2 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- control group: individuals without sarcopenia
- sarcopenic group: individuals with sarcopenia

SUMMARY:
The aim of this observational study is to reveal the effect of sarcopenia on cervical proprioception, kinesiophobia and pressure pain threshold in geriatric individuals living in a nursing home. The main questions it aims to answer are as follows:

The presence of sarcopenia in geriatric individuals living in a nursing home is effective/not effective on cervical proprioception.

The presence of sarcopenia in geriatric individuals living in a nursing home is effective/not effective on kinesiophobia.

The presence of sarcopenia in geriatric individuals living in a nursing home is effective/not effective on pressure pain threshold.

As a result of the evaluations, we will obtain the answers to the above questions with the surveys and measurements conducted with the participants divided into two groups as control and sarcopenia groups.

DETAILED DESCRIPTION:
Aging, which is a physiological process, is a period that reduces or limits the activity level and functionality of individuals, making them socially, physically and emotionally dependent to different degrees. With increasing age, changes may occur in physiological, psychological, cognitive and social areas, while the individual's cognitive and functional capacity decreases, an increase in the incidence of chronic diseases is observed. In light of today's scientific, medical, technological and economic developments, the population of both our country and the world is increasing. The 'geriatric syndrome concept' that we encounter due to the increasing elderly population has brought with it a series of sub-concepts. The most important of these concepts is the concept of sarcopenia, which has been the subject of many studies in recent years. Sarcopenia is defined as a progressive and widespread loss of muscle mass, function and strength. The EWGSOP, known as the European Working Group on Sarcopenia in the Elderly, defined sarcopenia in 2010 as a syndrome characterized by progressive and widespread loss of skeletal muscle mass and function, associated with risks such as physical disability, poor quality of life and death.

Sarcopenia, which is the most common among geriatric syndromes, significantly affects the physical, social and psychological life of the individual, while visibly restricting daily life activities. The presence of sarcopenia increases the risk and duration of hospitalization due to the loss of strength, falls and fragility it brings, and significantly increases the cost of care. Determining the parameters affected by sarcopenia in the geriatric population is essential for the establishment of preventive treatment algorithms and providing clinicians with a comprehensive perspective on sarcopenia.

The first factor that the presence of sarcopenia can affect may be proprioception. It is thought that the impairments in proprioception may be due to a decrease in the dynamic response of muscle spindles and axonal atrophy leading to impaired processing of sensory information. The cervical region is especially critical in terms of proprioception. The suboccipital muscles in the cervical region contain a large number of mechanoreceptors for proprioception, and this region is defined as the main source of proprioceptive information. However, there is no study in the literature investigating the relationship between sarcopenia and cervical proprioception or the effect of sarcopenia on cervical proprioception.

Another issue that needs to be addressed in the presence of sarcopenia is kinesiophobia. In a study conducted in 2024, the relationship between sarcopenia risk and kinesiophobia in geriatric individuals was evaluated and it was observed that sarcopenia risk increased the risk of kinesiophobia.

Finally, another issue that we want to evaluate in the presence of sarcopenia is the pressure pain threshold. No study investigating the relationship between sarcopenia and pressure pain threshold was found in the literature.

In light of the above information, the aim of the current study is to reveal the effect of sarcopenia on cervical proprioception, kinesiophobia and pressure pain threshold in geriatric individuals living in a nursing home.

Purpose: To reveal the effect of sarcopenia on cervical proprioception, kinesiophobia and pressure pain threshold in geriatric individuals living in a nursing home.

The current study was planned as a prospective, controlled study at the Private Nevia Oran Nursing Home and Elderly Care Center.

Universe and sample of the study: The study will be conducted with the participation of individuals living in the Private Nevia Oran Nursing Home and Elderly Care Center located in the city center of Ankara.

Data collection: Data will be collected by the researcher using a face-to-face interview technique .

To determine the sarcopenia classification, hand grip strength will be measured with the Jamar hand dynamometer, and physical performance will be evaluated with the the 4 m walking test . Bioimpedance Analysis (BIA) and anthropometric measurement methods will be used to measure muscle mass. Based on the results obtained, individuals will be divided into 2 groups as those with sarcopenia and those without sarcopenia.

Those with no decrease in muscle mass, grip strength and muscle performance will form the asymptomatic control group, while those with decreased muscle mass, grip strength and/or performance will be included in the sarcopenic group (experimental group).

Joint position error test will be used to assess cervical proprioception. An algometer will be used to assess the pressure pain threshold. The kinesiophobia causes scale and pain catastrophizing scale will be used to assess fear of movement and pain catastrophizing.

ELIGIBILITY:
Inclusion Criteria:

* Being 65 years of age or older
* Receiving a score of 24 or higher, which is considered mentally healthy, according to the mini mental assessment
* Having at least 91 points or more according to the Barthel daily living activities index (being mildly dependent or completely independent)

Exclusion Criteria:

* Having a disability (such as limb, vision, hearing loss),
* Having a serious neurological, orthopedic or rheumatological disorder that may affect proprioception,
* Having uncontrolled hypertension/diabetes,
* Having pain in the spine and/or extremities,
* Having a psychiatric disease diagnosis.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Geriatric people who lives in a nursing home in Ankara called Nevia Oran nursing home
Sampling Method: Non-Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2025-04-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
Assessment of cervical proprioception | 0-8 months
  Cervical proprioception was assessed using joint position error test . While seated, the participant faced a board positioned 90 cm away at head level, consisting of concentric circles (40 cm diameter, 1-cm increments), and wore a cap with a mounted laser pointer The participant first aligned the laser with the central point to establish the neutral position, then-with eyes open-was guided through flexion, extension, right/left rotation, and right/left lateral flexion, returning to neutral after each movement. The same six movements were then actively performed with eyes closed . Six repetitions were completed for each direction, and the point at which the laser stopped was marked on the board after every trial . The mean of these points was calculated, and angular deviation from the target was determined using the arctan method based on the fixed distance to the board. A deviation of more than 4 degrees was considered to indicate impaired proprioception.
Assessment of kinesiophobia | 0-8 months
  Kinesiophobia was assessed using the Kinesiophobia Causes Scale (KCS) . Developed by Kocjan and Knapik, the scale identifies the biological and psychological sources of fear of movement and contributes to understanding the underlying causes of reduced motor activity. It comprises two domains: biological and psychological. The biological domain includes morphological factors, movement requirements, energy resources, biological drives, negative experiences, motor competence, and beliefs related to body care, while the psychological domain assesses factors such as confidence, self-efficacy, and social interaction that contribute to avoidance behavior . The Turkish validity and reliability study was conducted by Çayır et al. The greater this value in the range of 0-5, the more valid the person's level of kinesiophobia.
Assessment of pressure pain threshold | 0-8months
  A pressure algometer (Baseline Force Gauge Model 12-0304; Baseline, NY, USA) will be used to assess the pressure pain threshold. The patient will be seated, and pressure will be applied perpendicularly and bilaterally using the algometer to different points in the cervical region (2 cm lateral to the C2 and C7spinous processes, at the midpoint of the upper part of the trapezius muscle) at a rate of approximately 3 N/s over an area of 0.5 cm² . The participant will be asked to report the moment they first felt discomfort and the pressure value at this moment will be recorded as the "pressure pain threshold". A second measurement will be taken at each region after an interval, the average of the two measurements will be noted.

CONTACTS AND LOCATIONS:
Overall Officials: nagihan acet, assistant professor, Study Director — atılım üniversity
Locations (1):
- Nevia Oran Nursing Home, Ankara, çankaya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
only IPD used in the results
Supporting Information: CSR

REFERENCES:
- [Background] Coşkun-Çelik, E., Medulla spinalis yaralanmalı hastalardaki nöropatik ağrıya akupunktur benzeri TENS'in etkisi. Uzmanlık Tezi, 2005.
- [Background] Gürel, Ö., Değişik muskuloskeletal sistem hastalıklarının basınç ağrı eşiği üzerine etkisi. Uzmanlık Tezi, Haydarpaşa Numune Eğitim ve Araştırma Hastanesi Fiziksel Tıp ve Rehabilitasyon Kliniği, İstanbul, 2009.
- [Background] Mekanizmaları, E.S.A., Ağrı Sendromları ve Tedavisi 2. baskı. İstanbul: Gizben Matbaacılık, 2003: p. 33-42.261.
- [Background] Düzel, V., Hemşire ve hastaların postoperatif ağrı değerlendirmelerinin karşılaştırılması. Çukurova Üniversitesi Sağlık Bilimleri Enstitüsü Yüksek Lisans Tezi. Adana, 2008.
- [Background] Akyol, B., Üst ekstremite ve bel ağrı tanısı konulmuş sedanter kadınlarda kalistenik egzersizlerin ağrı eşiği üzerine etkisi. Yayımlanmamış doktora tezi), İnönü Üniversitesi, Malatya, 2014.
- [Background] Wheeler CHB, Williams ACC, Morley SJ. Meta-analysis of the psychometric properties of the Pain Catastrophizing Scale and associations with participant characteristics. Pain. 2019 Sep;160(9):1946-1953. doi: 10.1097/j.pain.0000000000001494. PMID 30694929
- [Background] Osman A, Barrios FX, Kopper BA, Hauptmann W, Jones J, O'Neill E. Factor structure, reliability, and validity of the Pain Catastrophizing Scale. J Behav Med. 1997 Dec;20(6):589-605. doi: 10.1023/a:1025570508954. PMID 9429990
- [Background] Ugurlu, M., et al., Validity of Turkish form of Pain Catastrophizing Scale and modeling of the relationship between pain-related disability with pain intensity, cognitive, and emotional factors. Psychiatry and Clinical Psychopharmacology, 2017. 27(2): p. 189-196.
- [Background] Sullivan, M.J., S.R. Bishop, and J. Pivik, The pain catastrophizing scale: development and validation. Psychological assessment, 1995. 7(4): p. 524.,
- [Background] Kocjan, J. and A. Knapik, Barriers of physical activity (kinesiophobia) in patients subjected to cardiac rehabilitation. Baltic journal of health and physical activity, 2014. 6(4): p. 7.
- [Background] Knapik A, Saulicz E, Gnat R. Kinesiophobia - introducing a new diagnostic tool. J Hum Kinet. 2011 Jun;28:25-31. doi: 10.2478/v10078-011-0019-8. Epub 2011 Jul 4. PMID 23487514
- [Background] Çayır, M., N.A. Durutürk, and M.A. Tekindal, Kinezyofobi Nedenleri Ölçeği'nin Türkçe uyarlamasının geçerlik ve güvenirliği. Journal of Exercise Therapy and Rehabilitation, 2020. 7(1): p. 64-73.
- [Background] GENÇ, F.Z. and N. BİLGİLİ, Huzurevinde Yaşayan Yaşlılarda Kinezyofobi ve İlişkili Faktörlerin Değerlendirilmesi. Balıkesir Sağlık Bilimleri Dergisi, 2023. 12(2): p. 294-303.
- [Background] Benjaminse A, Sell TC, Abt JP, House AJ, Lephart SM. Reliability and precision of hip proprioception methods in healthy individuals. Clin J Sport Med. 2009 Nov;19(6):457-63. doi: 10.1097/JSM.0b013e3181bcb155. PMID 19898072
- [Background] Ager AL, Borms D, Deschepper L, Dhooghe R, Dijkhuis J, Roy JS, Cools A. Proprioception: How is it affected by shoulder pain? A systematic review. J Hand Ther. 2020 Oct-Dec;33(4):507-516. doi: 10.1016/j.jht.2019.06.002. Epub 2019 Aug 31. PMID 31481340
- [Background] Woollacott MH, Shumway-Cook A, Nashner LM. Aging and posture control: changes in sensory organization and muscular coordination. Int J Aging Hum Dev. 1986;23(2):97-114. doi: 10.2190/VXN3-N3RT-54JB-X16X. PMID 3557634
- [Background] Ferlinc A, Fabiani E, Velnar T, Gradisnik L. The Importance and Role of Proprioception in the Elderly: a Short Review. Mater Sociomed. 2019 Sep;31(3):219-221. doi: 10.5455/msm.2019.31.219-221. PMID 31762707
- [Background] Kristjansson E, Treleaven J. Sensorimotor function and dizziness in neck pain: implications for assessment and management. J Orthop Sports Phys Ther. 2009 May;39(5):364-77. doi: 10.2519/jospt.2009.2834. PMID 19411769
- [Background] Bahat G, Tufan A, Kilic C, Karan MA, Cruz-Jentoft AJ. Prevalence of sarcopenia and its components in community-dwelling outpatient older adults and their relation with functionality. Aging Male. 2020 Dec;23(5):424-430. doi: 10.1080/13685538.2018.1511976. Epub 2018 Oct 5. PMID 30290756
- [Background] Bahat G, Tufan A, Kilic C, Aydin T, Akpinar TS, Kose M, Erten N, Karan MA, Cruz-Jentoft AJ. Cut-off points for height, weight and body mass index adjusted bioimpedance analysis measurements of muscle mass with use of different threshold definitions. Aging Male. 2020 Dec;23(5):382-387. doi: 10.1080/13685538.2018.1499081. Epub 2018 Sep 29. PMID 30269625
- [Background] Janssen I, Heymsfield SB, Baumgartner RN, Ross R. Estimation of skeletal muscle mass by bioelectrical impedance analysis. J Appl Physiol (1985). 2000 Aug;89(2):465-71. doi: 10.1152/jappl.2000.89.2.465. PMID 10926627
- [Background] Ellis KJ, Bell SJ, Chertow GM, Chumlea WC, Knox TA, Kotler DP, Lukaski HC, Schoeller DA. Bioelectrical impedance methods in clinical research: a follow-up to the NIH Technology Assessment Conference. Nutrition. 1999 Nov-Dec;15(11-12):874-80. doi: 10.1016/s0899-9007(99)00147-1. PMID 10575664
- [Background] Bahat G, Tufan A, Tufan F, Kilic C, Akpinar TS, Kose M, Erten N, Karan MA, Cruz-Jentoft AJ. Cut-off points to identify sarcopenia according to European Working Group on Sarcopenia in Older People (EWGSOP) definition. Clin Nutr. 2016 Dec;35(6):1557-1563. doi: 10.1016/j.clnu.2016.02.002. Epub 2016 Feb 11. PMID 26922142
- [Background] Dodds R, Sayer AA. Sarcopenia. Arq Bras Endocrinol Metabol. 2014 Jul;58(5):464-9. doi: 10.1590/0004-273000000. PMID 25166036
- [Background] Testa G, Vescio A, Zuccala D, Petrantoni V, Amico M, Russo GI, Sessa G, Pavone V. Diagnosis, Treatment and Prevention of Sarcopenia in Hip Fractured Patients: Where We Are and Where We Are Going: A Systematic Review. J Clin Med. 2020 Sep 17;9(9):2997. doi: 10.3390/jcm9092997. PMID 32957453
- [Background] Cruz-Jentoft AJ, Bahat G, Bauer J, Boirie Y, Bruyere O, Cederholm T, Cooper C, Landi F, Rolland Y, Sayer AA, Schneider SM, Sieber CC, Topinkova E, Vandewoude M, Visser M, Zamboni M; Writing Group for the European Working Group on Sarcopenia in Older People 2 (EWGSOP2), and the Extended Group for EWGSOP2. Sarcopenia: revised European consensus on definition and diagnosis. Age Ageing. 2019 Jan 1;48(1):16-31. doi: 10.1093/ageing/afy169. PMID 30312372
- [Background] Yee XS, Ng YS, Allen JC, Latib A, Tay EL, Abu Bakar HM, Ho CYJ, Koh WCC, Kwek HHT, Tay L. Performance on sit-to-stand tests in relation to measures of functional fitness and sarcopenia diagnosis in community-dwelling older adults. Eur Rev Aging Phys Act. 2021 Jan 8;18(1):1. doi: 10.1186/s11556-020-00255-5. PMID 33419399
- [Background] Yoshiko A, Ogawa M, Shimizu K, Radaelli R, Neske R, Maeda H, Maeda K, Teodoro J, Tanaka N, Pinto RS, Akima H. Chair sit-to-stand performance is associated with diagnostic features of sarcopenia in older men and women. Arch Gerontol Geriatr. 2021 Sep-Oct;96:104463. doi: 10.1016/j.archger.2021.104463. Epub 2021 Jun 14. PMID 34218157
- [Background] HALİL, M., Z. ÜLGER, and S. ARIOĞLU, Sarkopeniye yaklaşım. Hacettepe Tıp Dergisi. 42. S: 123-132. 2011.
- [Background] Fielding RA, Vellas B, Evans WJ, Bhasin S, Morley JE, Newman AB, Abellan van Kan G, Andrieu S, Bauer J, Breuille D, Cederholm T, Chandler J, De Meynard C, Donini L, Harris T, Kannt A, Keime Guibert F, Onder G, Papanicolaou D, Rolland Y, Rooks D, Sieber C, Souhami E, Verlaan S, Zamboni M. Sarcopenia: an undiagnosed condition in older adults. Current consensus definition: prevalence, etiology, and consequences. International working group on sarcopenia. J Am Med Dir Assoc. 2011 May;12(4):249-56. doi: 10.1016/j.jamda.2011.01.003. Epub 2011 Mar 4. PMID 21527165
- [Background] Cruz-Jentoft AJ, Sayer AA. Sarcopenia. Lancet. 2019 Jun 29;393(10191):2636-2646. doi: 10.1016/S0140-6736(19)31138-9. Epub 2019 Jun 3. PMID 31171417
- [Background] Telli, H. and Ç. Özdemir, The Effects of Sarcopenia and Fracture Risk on Kinesiophobia, Fear of Falling, Fall Risk and Quality of Life in Geriatric Individuals. Turk J Osteoporos, 2024. 30(2): p. 75-88.
- [Background] Kulkarni V, Chandy MJ, Babu KS. Quantitative study of muscle spindles in suboccipital muscles of human foetuses. Neurol India. 2001 Dec;49(4):355-9. PMID 11799407
- [Background] Humphreys BK. Cervical outcome measures: testing for postural stability and balance. J Manipulative Physiol Ther. 2008 Sep;31(7):540-6. doi: 10.1016/j.jmpt.2008.08.007. PMID 18804005
- [Background] Ribeiro, F. and J. Oliveira, Aging effects on joint proprioception: the role of physical activity in proprioception preservation. European review of aging and physical activity, 2007. 4(2): p. 71-76.
- [Background] Cawthon PM, Lui LY, Taylor BC, McCulloch CE, Cauley JA, Lapidus J, Orwoll E, Ensrud KE. Clinical Definitions of Sarcopenia and Risk of Hospitalization in Community-Dwelling Older Men: The Osteoporotic Fractures in Men Study. J Gerontol A Biol Sci Med Sci. 2017 Oct 1;72(10):1383-1389. doi: 10.1093/gerona/glw327. PMID 28329087
- [Background] Steffl M, Bohannon RW, Sontakova L, Tufano JJ, Shiells K, Holmerova I. Relationship between sarcopenia and physical activity in older people: a systematic review and meta-analysis. Clin Interv Aging. 2017 May 17;12:835-845. doi: 10.2147/CIA.S132940. eCollection 2017. PMID 28553092
- [Background] Schaap LA, van Schoor NM, Lips P, Visser M. Associations of Sarcopenia Definitions, and Their Components, With the Incidence of Recurrent Falling and Fractures: The Longitudinal Aging Study Amsterdam. J Gerontol A Biol Sci Med Sci. 2018 Aug 10;73(9):1199-1204. doi: 10.1093/gerona/glx245. PMID 29300839
- [Background] Dos Santos L, Cyrino ES, Antunes M, Santos DA, Sardinha LB. Sarcopenia and physical independence in older adults: the independent and synergic role of muscle mass and muscle function. J Cachexia Sarcopenia Muscle. 2017 Apr;8(2):245-250. doi: 10.1002/jcsm.12160. Epub 2016 Nov 8. PMID 27897417
- [Background] Bischoff-Ferrari HA, Orav JE, Kanis JA, Rizzoli R, Schlogl M, Staehelin HB, Willett WC, Dawson-Hughes B. Comparative performance of current definitions of sarcopenia against the prospective incidence of falls among community-dwelling seniors age 65 and older. Osteoporos Int. 2015 Dec;26(12):2793-802. doi: 10.1007/s00198-015-3194-y. Epub 2015 Jun 12. PMID 26068298
- [Background] Cruz-Jentoft AJ, Baeyens JP, Bauer JM, Boirie Y, Cederholm T, Landi F, Martin FC, Michel JP, Rolland Y, Schneider SM, Topinkova E, Vandewoude M, Zamboni M; European Working Group on Sarcopenia in Older People. Sarcopenia: European consensus on definition and diagnosis: Report of the European Working Group on Sarcopenia in Older People. Age Ageing. 2010 Jul;39(4):412-23. doi: 10.1093/ageing/afq034. Epub 2010 Apr 13. PMID 20392703
- [Background] Derya, K., et al., Geriatri poliklinik olgularında geriatrik sendromlar: 1048 olgunun analizi. Ege Tıp Dergisi, 2018. 57(1): p. 31-35.
- [Background] Carlson C, Merel SE, Yukawa M. Geriatric syndromes and geriatric assessment for the generalist. Med Clin North Am. 2015 Mar;99(2):263-79. doi: 10.1016/j.mcna.2014.11.003. Epub 2015 Jan 10. PMID 25700583
- [Background] Buz, S., Yaşlı bireylere yönelik yaş ayrımcılığı. Elektronik Sosyal Bilimler Dergisi, 2015. 14(53).
- [Background] Beğer, T. and H. Yavuzer, Yaşlılık ve yaşlılık epidemiyolojisi. Klinik gelişim, 2012. 25(3): p. 1-3.
- See also: Related Info — https://scholar.google.com/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/